CLINICAL TRIAL: NCT03074968
Title: Effect of Benzydamine Hydrochloride to Postoperative Sore Throat in Pediatric Patients: a Randomized Controlled Trial
Brief Title: Effect of Benzydamine Hydrochloride to Postoperative Sore Throat in Pediatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H1612-061-813
Record Dates: First submitted 2017-02-26; First posted 2017-03-09 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Intubation Complication
MeSH Terms: interventions — Benzydamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (Placebo Comparator): normal saline
  Interventions: Drug: Normal saline
- benzydamine hydrochloride (Active Comparator): Benzydamine Hydrochloride
  Interventions: Drug: Benzydamine Hydrochloride

INTERVENTIONS:
Drug: Benzydamine Hydrochloride — Benzydamine Hydrochloride application
  Other Names: difflam
  Arms: benzydamine hydrochloride
Drug: Normal saline — normal saline application
  Other Names: ns
  Arms: control

SUMMARY:
This study is designed to examine the effect of benzydamine hydrochloride to postoperative sore throat in pediatric patients. We will spray benzydmaine hydrochloride or normal saline at oral cavity and the tip of endotracheal tube, than compare the prevalence of postoperative sore throat using smartphone application in pediatric patients.

DETAILED DESCRIPTION:
1. postoperative sore throat incidence (over 2) 1; no, 2;mild, 3;moderate, 4;severe
2. scoring of pain with smartphone application (kids pain scale)
3. incidence of use of rescue pain killer

ELIGIBILITY:
Inclusion Criteria:

* general anesthesia
* intubation require

Exclusion Criteria:

* recent upper airway infection
* could not express the pain

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 142 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
pain | 30 minutes in postanesthetic care unit
  application based pain score

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, Principal Investigator — Seoul National University
Locations (1):
- SNUH, Seoul, Jongro Gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yhim HB, Yoon SH, Jang YE, Lee JH, Kim EH, Kim JT, Kim HS. Effects of benzydamine hydrochloride on postoperative sore throat after extubation in children: a randomized controlled trial. BMC Anesthesiol. 2020 Apr 4;20(1):77. doi: 10.1186/s12871-020-00995-y. PMID 32247315